CLINICAL TRIAL: NCT06432452
Title: Efficacy of Endothelin Receptor Antagonism in Treatment of Coronary Artery Spasm: a Randomized Controlled Clinical Trial
Brief Title: Efficacy of Endothelin Receptor Antagonism in Coronary Artery Spasm
Acronym: EDIT-CAS
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: UMC Utrecht (Other); Catharina Ziekenhuis Eindhoven (Other); Maasstad Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 114746
Record Dates: First submitted 2024-05-10; First posted 2024-05-29 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Coronary Spasm
Keywords: epicardial spasm; endothelin receptor antagonism; angina
MeSH Terms: conditions — Angina Pectoris, Variant; Angina Pectoris | interventions — Endothelin Receptor Antagonists; Bosentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bosentan (Experimental): Bosentan 62.5 mg twice daily Uptitrated to 125mg twice daily if tolerated after 4 weeks Total 10 weeks
  Interventions: Drug: Endothelin Receptor Antagonist
- Placebo (Placebo Comparator): Placebo 62.5 mg twice daily Uptitrated to 125mg twice daily if tolerated after 4 weeks Total 10 weeks
  Interventions: Other: Placebo control

INTERVENTIONS:
Drug: Endothelin Receptor Antagonist — Oral capsules twice daily
  Other Names: Bosentan
  Arms: Bosentan
Other: Placebo control — Oral capsules twice daily
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The goal of this randomized clinical trial is to assess if adjunctive bosentan therapy, in comparison to placebo, can reduce the rate of epicardial vasospasm at follow-up spasm provocation CFT (fuCFT) in patients with previously proven epicardial vasospasm on acetylcholine reactivity testing (at index CFT) and ongoing angina(-like) complaints.

Participants will

* Use either endothelin receptor antagonist or placebo for 10 weeks
* Undergo follow-up acetylcholine spasm provocation test after 10 weeks
* Answer online questionnaires on angina and quality of life

ELIGIBILITY:
Inclusion Criteria:

1. Definitive diagnosis of epicardial vasospasm on maximal acetylcholine dose of 100µg (at iCFT)
2. At least 18 years of age
3. On optimal regular care ( current or previous treatment with at least 2 daily anti-anginal medicines i.e. nitrate and calcium channel blocker
4. Continuing episodes of angina(-like) complaints at least once weekly despite 3.
5. Signed online informed consent for participation in NL-CFT registry (the Netherlands Registry of invasive coronary vasomotor function testing), or willing to co-sign for registry at time of inclusion in EDIT-CAS
6. Written informed consent for EDIT-CAS

Exclusion Criteria:

1. Systolic blood pressure (SBP) <85 mmHg measured at Visit 1
2. Significant hepatic impairment at time of iCFT lab (ASAT/ALAT >3x upper limit of normal (ULN)) or history of liver cirrhosis (Child-Pugh 7-15)
3. Severe anemia (Hb<6.0mmol/L) without identified cause at time of inclusion
4. Patients with limited life expectancy (<1 year)
5. Participation in another randomized clinical study with an use of an Investigational Medicinal Product (IMP) up to one month prior to enrolment.
6. Pregnancy, active desire to become pregnant or unwilling to take adequate* contraceptive measures when of child bearing potential for the duration of 6 months (active medication period + 3 months safety).
7. Known heart failure with reduced ejection fraction<35%
8. Known pulmonary hypertension of any type
9. Potentially dangerous interaction due to the use of another CYP3A4 or CYP2C9 substrate (e.g. ciclosporin A, glibenclamide, fluconazole, rifampicin, tacrolimus/sirolimus, lopinavir/ritonavir)
10. Repeat spasm provocation test deemed unsafe (e.g. allergic reaction at iCFT)

    * Adequate in this case meaning if on hormonal contraceptives, additional measures to be taken (e.g. condom).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Successful treatment | 10 weeks
  On repeat invasive spasm provocation according to Coronary Vasomotor Disorders International Study Group (COVADIS) criteria. Successful treatment is defined as absence of epicardial vasospasm according to COVADIS criteria during repeat spasm provocation test at 10 weeks.

SECONDARY OUTCOMES:
Improvement of anginal complaints | 10 weeks
  As measured with Seattle Angina Questionnaire (SAQ) summary score and change from baseline to follow-up. Score can range from 0-100, with higher scores indicating better health status.

OTHER OUTCOMES:
Improvement of quality of life | 10 weeks
  Measured with EuroQol 5 Dimensions (EQ5D) and separate SAQ domains. Scores can range from 0-100, with higher scores indicating better health status.
Microvascular spasm | 10 weeks
  The rate of occurence of microvascular spasm according to COVADIS criteria at fuCFT
Endothelin levels at baseline | 10 weeks
  Circulating endothelin-1 plasma levels in peripheral blood drawn at visit 1.
Change in spasm provocation reactivity | 10 weeks
  Any deterioration or improvement according to prespecified outcomes measured by repeated spasm provocation test. If a higher dose of acetylcholine is needed to induce epicardial spasm for example, this change will be documented. If microvascular spasm can, but epicardial can not be provoked, this will be documented. The incidence of these changes will be analyzed.
Incidence of liver panel disturbances | 10 weeks
  Assessed by means of repeat laboratory analysis
Incidence of hypotension | 10 weeks
  Assessed by means of repeat blood pressure measurements
Incidence of MACE | 10 weeks
  Assessed by (S)AE reporting, during all follow-up contacts
Rate of study drug discontinuation / study withdrawal. | 10 weeks
  Assessed and captured at every follow-up contact moment.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Damman, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (4):
- Netherlands (4):
  - Catharina Ziekenhuis, Eindhoven, North Brabant
  - Maasstad Hospital, Rotterdam, South Holland
  - RadboudUMC, Nijmegen
  - UMC Utrecht, Utrecht

REFERENCES:
- [Derived] Crooijmans C, Jansen T, van de Hoef T, Paradies V, de Vos A, Yosofi B, Cetinyurek-Yavuz A, den Ruijter H, Beijk M, Meuwissen M, van Royen N, Elias-Smale S, Dimitriu-Leen A, Damman P; for NL-CFT. Design and rationale of the efficacy of endothelin receptor antagonism in treatment of coronary artery spasm: a randomized controlled trial (EDIT-CAS). Am Heart J. 2025 Oct;288:140-148. doi: 10.1016/j.ahj.2025.04.022. Epub 2025 Apr 22. PMID 40274007